CLINICAL TRIAL: NCT03237975
Title: A Strengths-based Intervention Based on Salutogenic Theory to Promote Sense of Coherence and Self-care of Elderly People With Type 2 Diabetes
Brief Title: BEYO Project to Promote Sense of Coherence and Self-care of Elderly People With Type 2 Diabetes
Acronym: BEYO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lei Yang, Graduate Assistant, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BEYO Project-LYCUHK
Record Dates: First submitted 2017-07-24; First posted 2017-08-03 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-07

CONDITIONS: Diabetes Mellitus, Type 2; Sense of Coherence; Self Care; Strengths-based Intervention
Keywords: type 2 diabetes; sense of coherence; self-care; strengths-based intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Participants were assigned to two groups in parallel for the duration of the study. One group received usual care for diabetes patients. One group received strengths-based intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Be the Expert for Your Own (BEYO) (Experimental): BEYO is a group-based consultation project. Each group contains 1 facilitator, 1 assistant and 8 elderly patients. 5 weekly sessions are provided to let patients receive health knowledge, discuss problems and experiences, explore available resources and build up goals and solutions. Each session lasts for 40 minutes. Session 1 aims to build social network among group members and introduce group goals and tasks. Session 2-4 covers six topics: (i) healthy dietary, (ii) exercise and activity, (iii) taking medication, (iv) blood glucose monitoring, (v) reducing risks for complication, (vi) healthy coping with mental stress. Session 5 aims to review the process, summarize effective solutions, and set up plans for the future.
  Interventions: Behavioral: Be the Expert for Your Own (BEYO)
- Routine health education (Active Comparator): To neutralize the effect of extra attention from the facilitator, participants in control group will receive routine health education on topics related to type 2 diabetes. Contents for the routine education will be based on the national guideline of basic public health service for diabetes and specific implementation protocols in each community. Participants in control group will receive 5-weekly education packet at the same time with participants in intervention group. The patients will not be given any strengths-based information, but they are free to discuss their disease status with nurses or physicians at their regular follow-up appointments.
  Interventions: Other: Routine health education

INTERVENTIONS:
Behavioral: Be the Expert for Your Own (BEYO) — The BEYO program is structured adopting solution focused therapy (SFT). The basic principles for SFT are focusing on positive change and establishing groups driven by goals rather than problems. Solutions are generated through searching for strengths, skills, resources that working in clients' lives.
  The common flow for structured sessions contains 7 steps: 1) Health education; 2) Discuss self-care experience and identify deficit; 3) Describe exceptions; 4) Identify the strengths; 5) Miracle question and scaling; 6) Establish the solution; 7) Action plan.
  Arms: Be the Expert for Your Own (BEYO)
Other: Routine health education — The control group will receive routine health education.
  Arms: Routine health education

SUMMARY:
1. Objectives of the Project

   The BEYO project is designed based on the middle range theory of self-care of chronic illness and salutogenic theory. The aim of this project is to facilitate self-care behaviours of community-dwelling elderly patients with type 2 diabetes through promoting SOC, and accordingly improve their health outcomes, including promoting quality of life and reducing diabetes-related emotional distress.
2. Content of the Project

BEYO is a group-based consultation project. Each group contains 1 facilitator, 1 assistant and 8 elderly patients. 5 weekly sessions are provided to let patients receive health knowledge, discuss problems and experiences, explore available resources and build up goals and solutions. Each session lasts for 40 minutes. Session 1 aims to build social network among group members and introduce group goals and tasks. Session 2-4 covers six topics based on the Chinese guideline for type 2 diabetes released by Chinese diabetes society: (i) healthy dietary, (ii) exercise and activity, (iii) taking medication, (iv) blood glucose monitoring, (v) reducing risks for complication, (vi) healthy coping with mental stress. These middle sessions execute a common session flow to construct an action plan utilizing patients' resources and strengths to achieve the client-centered goal. Session 5 aims to review the process, summarize effective solutions, and set up plans for the future. One-week, one-month and three-month telephone follow-ups are delivered to help patients solve problems encountered during implementing the action plan and evaluate their self-care, SOC and other health outcomes.

DETAILED DESCRIPTION:
1. Overall aims The aim of this study is to develop and evaluate the effects of a strengths-based group intervention called Be the Expert for Your Own (BEYO) among elderly patients with type 2 diabetes to facilitate their SOC and self-care, and accordingly improve their health outcomes.
2. Study Design This study is designed to be a mixed method research incorporating both quantitative and qualitative components. A two-arm randomized controlled trial (RCT) will be conducted to assess the effects of a strengths-based group intervention compared with routine health education on SOC and self-care of elderly people with type 2 diabetes. The theoretical framework for BEYO program is based on salutogenic theory proposed by Antonovsky (1987). Qualitative study will be conducted at the end of the program to explore patients' experience about BEYO and the mechanism through which BEYO can facilitate self-care, in terms of what component and how.

2. Be the Expert for Your Own (BEYO) program

1. Overview The BEYO protocol consists of 5 structured sessions among intervention facilitator and 8 type 2 diabetes patients.The common flow for structured sessions contains 7 steps. Rationale and aims for designing each step are described as follows.

   Step 1 - "Health education" As supported by the middle range theory and results from integrated review, knowledge acquisition is essential among patients with chronic disease to perform reflective, sufficient and reasoned self-care actions with a pattern. This step aims to equip patients with basic knowledge and essential skills to manage their disease.

   Step 2 - "Discuss self-care experience and identify deficit" This step aims to collect basic information about clients' experience of performing self-care in each specific area and identify major problems they encounter in this process. This step facilitates information exchange and experience sharing among clients and provides reference for intervention facilitator about clients' basic situation. Besides, giving enough opportunity to describe the problem makes it easier to redirect the conversation later if attendees restart talking about the problem.

   Step 3 - "Describe exceptions" One of the central beliefs for SFT is that there are always exceptions to problems. There are always times and situations when the problem occurs less or when the client feels like successfully managing even a slight part of the problem. After identifying self-care deficit, clients are asked to describe these exceptional times in this step to help them find out skills, resources, and strengths at their disposal. The close attention for exceptions improves clients' sense of self-mastery and their ability to plan further steps.

   Step 4 - "Identify the strengths" On the basis of review and analysis for exceptions, it is the right time to list out and summarize clients' strengths revealed in these exceptions. This step lays a foundation for establishing solutions later, for that detected strengths can be amplified and repeated to ultimately dismantle the problem.

   Step 5 - "Miracle question and scaling" The miracle question is a common tool in SFT as a way to build clear, client-centered and practical goals. Scaling questions help to break the goal down into small manageable steps that can be carried out in the short term. This step helps clients find out what they want to achieve through this program. Setting the goal by themselves facilitates an empowering and optimistic experience for clients that promoting goal-focused thinking during the self-care process and highlighting their responsibility for the future actions.

   Step 6 - "Establish the solution" After exploring strengths and setting up the goal, this step aims to link strengths and goals together to establish the solution. As the basic principles for SFT is focusing on strengths rather than weakness, resources rather than deficits, the created solution is more concerned with achievement than with solving problems, with hoping not just coping. It helps clients move forward in their lives.

   Step 7 - "Action plan" As the final step, a structured action plan is generated to transform the solution into arranged tasks. The action plan guides the behaviors of the clients and tracks the progress of implementation.
2. The role of facilitator Different with the traditional teacher-centered didactic model, facilitators in BEYO program need to get out of the expert role and appreciate patients' capabilities from the aspect of truly human beings. Rather than being at the center of the group, the facilitator is a supporter to assist patients to identify what they want to achieve, to help them to think about strengths and resources during the group interactions, to build up solutions for their own situations and to make plans to reach the goal step by step.

   To build a hope-inducing relationship between the facilitator and clients has been emphasized as the context for practice to enhance the effectiveness of strengths-based techniques (Fischer, 1978). The foundation for a hope-inducing relationship includes empathy, genuineness and unconditional positive regard (Maluccio, 1979). To be empathy, facilitators need to perceive and communicate feelings of attendees with sensitivity, and think about the meaning of these feelings. Genuineness means that facilitators should be themselves in the helping process rather than presenting a professional facade. Unconditional positive regard asks facilitators to give positive feedback to every good change and to express the respect, acceptance, caring and concern for the client in a non-dominating way.
3. Objectives for each session Session 1 aims to build social network among group members and make clients feel welcome. Group goals and task will be introduced to gel the clients around the group.

   Session 2-4 execute a common session flow to finally construct an action plan to achieve the client-centered goal. Themes for the total 3 sessions respectively cover the six areas as mentioned earlier. Except session 2, all the other sessions will start with reinforcing the positive change happening since the last session.

   Session 5 aims to celebrate the achievement, review the process, summarize clients' strengths and effective solutions, and set up plans for the future.
4. Acceptability and feasibility evaluation Researchers will record numbers and proportions for recruitment, consent, attendance, and attrition rate. Duration of sessions and intervention activities will be recorded using field notes. The research team and the facilitator will discuss the delivery of the program and study progress every week.

The focus-group interview will be conducted at the end of the study to explore patients' experience and opinions about the content and process, and barriers and enablers to compliance with the intervention.

3. Subjects

3.1 Sampling and recruitment The group of elderly patients with type 2 diabetes living in Changsha, a city in central China, is selected as the study population. Multi-stage random sampling will be used to recruit community-dwelling participants. First, two of the five municipal districts of Changsha City based on present administrative system will be randomly selected. Second, detailed information including names and numbers of community health service centers belong to each district can be achieved through government official websites. Two community health service centers respectively belong to the two districts will be randomly selected. Third, based on national standards of public health services, all the community-dwelling patients with type 2 diabetes should be recorded in the electronic medical system charged by the department of chronic disease management in the community health service center. Random number table method will be used to select potential participants in each of the two communities, using this electronic system. No private information of type 2 diabetes patients will be retrieved except for their name, mailing address and contact number.

An information sheet will be sent as a letter from the research team to the potential participant followed by a telephone call two days later. The phone call is mainly designed to (i) further make sure if the referrals meet the inclusion criteria, such as age and time of diagnosis; (ii) discuss the information sheet and obtain verbal informed consent for the project, (iii) verbally deliver Abbreviated Mental Test (AMT) and the Summary of Diabetes Self-Care Activities measure (SDSCA) to make sure the participants have intact cognitive function and experience at least some degree of self-care deficit for diabetes.

3.2 Sample size calculation The significance level and the power are set at 5% and 80% respectively. The primary outcome is self-care of elderly patients with type 2 diabetes. However, based on the result of literature review, no previous studies used strengths-based intervention reported its effects on self-care. Based on the result of a meta-analysis assessing effects of group-based diabetes self-management education compared to routine treatment (Steinsbekk, Rygg, Lisulo, Rise, & Fretheim, 2012), the standardized mean difference for self-care skills was 0.55. Thus, a sample size of 53 in each group is enough to detect the difference in the means of self-care between two groups. Allowing for a dropout rate of 20%, a total of 132 participants will be required.

3.3 Randomization After obtaining the signed informed consent form and collecting the baseline data, patients will be randomly allocated to the intervention or control group, using a computerized permuted block randomization with concealment.

4. Data Collection Data collection will be commenced after receiving written informed consent voluntarily signed by participants. The baseline information (T0) will be collected before the randomization. After completing the intervention or control protocol, a follow-up data collection (T1) will be conducted immediately by a group of trained research assistants, who are blinded to the participants' group assignment and workshop attendance. Repeated data collection (T2) will take place at 3 months after the completion of the strength-based intervention by the same group of research assistants.

5. Data Analysis Plan Invalid questionnaire (questionnaire with obvious logic error, or with more than 20% unanswered questions) will be excluded before put into the database. SPSS version 22.0 will be used to process data. The level of statistical significance will be set at 0.05. Q-Q plot, Skewness and Kurtosis will be used to examine the normality of continuous data. Descriptive statistics will be used to summarize the demographic characteristics, health status and patient-centered outcomes. The effectiveness of the intervention will be assessed based on the intention-to-treat (ITT) principle. The generalized estimating equation (GEE) model will be used to estimate the intervention effect over time. Hierarchical multiple regression analysis will be conducted to examine the mediating effect of sense of coherence.

ELIGIBILITY:
Inclusion Criteria:

1. A medical diagnosis of type 2 diabetes according to diagnostic criteria recommended by WHO (2006);
2. Older than aged 60 years;
3. Diagnosed with diabetes at least six months before the intervention;
4. Residing in the community, able to read and communicate in Chinese;
5. Having intact cognitive function as indicated by the Abbreviated Mental Test of score >=6;
6. Having some degree of self-care deficit as indicated by the Chinese version of SDSCA of score <=23.

Exclusion Criteria:

1. Presence of serious mental problem or terminal illness;
2. Previously participated in similar programs;
3. Visual or audio impaired.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
the Chinese version of the Summary of Diabetes Self-Care Activities measure (SDSCA) | From the date of recruitment, until the date of randomization, up to 2 weeks
  SDSCA is a brief self-report measure for assessing levels of self-care across different components of the diabetes regimen. The new version revised by Toobert's team (2000) uses 11 items to include 6 aspects of diabetes regimen: general diet, specific diet, exercise, blood-glucose testing, foot care, and smoking.
Short form of the sense of coherence questionnaire (SOC-13) | From the date of recruitment, until the date of randomization, up to 2 weeks
  The SOC questionnaire was developed by Antonovsky (1987) to measure three components of sense of coherence: comprehensibility, manageability and meaningfulness.
the Chinese version of the Summary of Diabetes Self-Care Activities measure (SDSCA) | 5 weeks after the project started
  SDSCA is a brief self-report measure for assessing levels of self-care across different components of the diabetes regimen. The new version revised by Toobert's team (2000) uses 11 items to include 6 aspects of diabetes regimen: general diet, specific diet, exercise, blood-glucose testing, foot care, and smoking.
Short form of the sense of coherence questionnaire (SOC-13) | 5 weeks after the project started
  The SOC questionnaire was developed by Antonovsky (1987) to measure three components of sense of coherence: comprehensibility, manageability and meaningfulness.
the Chinese version of the Summary of Diabetes Self-Care Activities measure (SDSCA) | 3-month after the project ended
  SDSCA is a brief self-report measure for assessing levels of self-care across different components of the diabetes regimen. The new version revised by Toobert's team (2000) uses 11 items to include 6 aspects of diabetes regimen: general diet, specific diet, exercise, blood-glucose testing, foot care, and smoking.
Short form of the sense of coherence questionnaire (SOC-13) | 3-month after the project ended
  The SOC questionnaire was developed by Antonovsky (1987) to measure three components of sense of coherence: comprehensibility, manageability and meaningfulness.

SECONDARY OUTCOMES:
the Chinese version of the Audit of Diabetes Dependent Quality of Life (CN-ADDQoL) | From the date of recruitment, until the date of randomization, up to 2 weeks; 5 weeks after the project started; 3-month after the project ended
  The ADDQoL is a diabetes-specific health related quality of life instrument (Bradley et al., 1999) assessed perceived impact of diabetes on 19 life domains containing physical functioning, symptoms, psychological well-being, social well-being, role activities and personal construct.
Diabetes Distress Scale (DDS) | From the date of recruitment, until the date of randomization, up to 2 weeks; 5 weeks after the project started; 3-month after the project ended
  The DDS is developed by Polonsky et al (2005) to assess diabetes-related emotional distress. DDS contains 17 items to cover 4 dimensions: emotional burden, physician-related distress, regimen-related distress, and diabetes-related interpersonal distress.
Diabetes Self-Efficacy Scale (DSES) | From the date of recruitment, until the date of randomization, up to 2 weeks; 5 weeks after the project started, 3-month after the project ended
  DSES was developed by Stanford Patient Education Research Center (Lorig et al., 2009), including 8 items to assess patients' confidence in areas including dietary, exercise and symptom management.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Lei, Principal Investigator — Chinese University of Hong Kong
Locations (2):
- China (2):
  - He Xinyuan Community Health Care Center, Changsha, Hunan
  - Yannong Neighborhood Health Care Clinics, Changsha, Hunan